CLINICAL TRIAL: NCT03425942
Title: Internet Administered CBT for Insomnia Comorbid With Chronic Pain Compared to Applied Relaxation Techniques - A Randomized Controlled Trial
Brief Title: Internet Administered CBT for Insomnia Comorbid With Chronic Pain
Acronym: SoV-studien
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Linkoeping University (Other Government)
Responsible Party: Principal Investigator, Bjorn Gerdle, Professor, Linkoeping University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: LIU-002
Record Dates: First submitted 2018-01-24; First posted 2018-02-08 (Actual); Last update posted 2021-01-11 (Actual); Status verified 2021-01

CONDITIONS: Insomnia Due to Medical Condition; Chronic Pain
Keywords: Cognitive Behavioral Therapy; Applied Relaxation Techniques; Internet treatment
MeSH Terms: conditions — Chronic Pain

STUDY DESIGN:
Who Masked: Participant
Masking Description: Participants in both the experiment condition and the active control group were told that they received one of two active treatments in a comparative study.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Internet CBT for insomnia (Experimental): The intervention consists of Internet-based Cognitive Behavioral Therapy for insomnia (ICBT-i) (the main components are sleep restriction and stimulus control) for five consecutive weeks.
  Interventions: Behavioral: Internet Cognitive Behavioral Therapy for insomnia (ICBT-i)
- Internet ART for insomnia (Active Comparator): The intervention consists of internet-based applied relaxation exercises/techniques (ART) (different and commonly used) for five consecutive weeks.The acronyme for this intervention is (IART-i).
  Interventions: Behavioral: Internet Applied Relaxation Techniques (IART-i)

INTERVENTIONS:
Behavioral: Internet Cognitive Behavioral Therapy for insomnia (ICBT-i) — This intervention lasts for five weeks. The intervention is internet-based and mainly consists of the most potent CBT technics i.e. sleep restriction and stimulus control. Weekly feedback is provided by master students supervised by clinical psychologists.
  Arms: Internet CBT for insomnia
Behavioral: Internet Applied Relaxation Techniques (IART-i) — This intervention lasts for five weeks. The intervention is internet-based and consists of different common applied relaxation exercises and treatments. Weekly feedback is provided by master students supervised by clinical psychologists.
  Arms: Internet ART for insomnia

SUMMARY:
Cognitive behavioural therapy (CBT), that is designed to be short, concise and user friendly is compared to applied relaxation techniques as treatment for insomnia comorbid with chronic pain. Both treatments are administered via internet and participants are randomized to ether treatment arm.

DETAILED DESCRIPTION:
Internet treatment with therapist support means that measurements are collected through the Internet. Participants are recruited from a specialized pain clinic for chronic pain. All patients with sleep complaints (Insomnia Severity Index > 14) at their first visit through 2016-01-01 to 2017-07-31 are asked for participation via mail. Volunteers sign informed consent and undergo a online screening. If matching the inclusion criteria, they are contacted for a telephone interview. Subjects are assessed according to the Diagnostic and Statistical Manual of Mental Disorders, Fifth Edition (DSM-5) criterion for insomnia disorder, M.I.N.I. (screening for psychiatric comorbidity) and the other inclusion/exclusion criteria. The treatment, that is designed to be short, concise and user friendly as it is meant to be usable as an adjunct treatment to other main interventions for chronic pain. The treatment lasts for five weeks and focuses on the most potent CBT technics for insomnia; sleep restriction and stimulus control.

Randomization is conducted by university staff not otherwise involved in this study. Participants have equal chance to be allocated to ether CBT or applied relaxation techniques (active controls). The relaxation treatment lasts for the same amount of time (five weeks) and is designed to require similar weekly effort. Both groups fill in sleep diaries every week and weekly feedback is provided by master students supervised by clinical psychologists.

The overall hypothesis is that CBT leads to greater symptom reduction (according to the Insomnia Severity Index) compared to applied relaxation techniques.

ELIGIBILITY:
Inclusion Criteria:

* Insomnia severity index (ISI) score > 14
* Chronic pain

Exclusion Criteria:

* Shift worker or employed as a driver, operator of dangerous equipment and such
* Sleep apnea, restless legs syndrome, narcolepsy, Myalgic Encephalomyelitis/Chronic Fatigue Syndrome (ME/CFS)
* Bipolar disorder, psychotic disorders, ongoing substance abuse
* Having received CBT for insomnia during the latest year
* Pregnancy
* Severe somatic disorder (such as ongoing cancer, severe neurological condition, insufficiently treated cardiac condition)
* Impaired movement to such a degree that going to bed or getting out of bed requires assistance
* Not being able read or wright in Swedish
* Not having an internet-connected computer, cellular phone or tablet

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 54 (Actual)
Dates: Start 2018-02-09 (Actual); Primary Completion 2019-05-07 (Actual); Study Completion 2019-05-14 (Actual)

PRIMARY OUTCOMES:
Insomnia Severity Index (ISI) | Change from baseline insomnia severity (ISI) at 6 months
  Measures degree of insomnia. Range 0-28 where a higher value indicates worse sleep.

SECONDARY OUTCOMES:
Sleep diary | Daily during treatment (five weeks).
  Basis for sleep latency, total sleep time, wake time after sleep onset and sleep efficiency.
The Karolinska Sleepiness Scale (KSS) | Change from baseline sleepiness (KSS) at 5 weeks
  Measures sleepiness on a single item numeric rating scale. Range 1-9, where a higher value indicates more sleepiness.
Patient Health Questionnaire (PHQ-9) | Change from baseline health (PHQ-9) at 6 months
  Measures depressive symptoms. Range 0-27, where a higher value indicates more depressive symptoms.
Generalised Anxiety Disorder 7-item scale (GAD-7) | Change from baseline anxiety (GAD-7) at 6 months
  Measures anxiety symptoms. Range 0-21 where a higher value indicates more anxiety.
Pain intensity (NRS) | Change from baseline pain intensity (NRS) at 6 months
  Eleven stepped numeric rating scale (NRS) for average pain last seven days. Higher values indicate higher pain intensity.
Pain Disability Index (PDI) | Change from baseline disability (PDI) at 6 months
  Quantifying pain related disability. Range 0-70 where a higher value indicates more disability.

OTHER OUTCOMES:
Pain spreading (PS) | Change from baseline pain spreading (PS) at 6 months
  Number of anatomical regions with pain out of 36 anatomical areas.
Negative Effects Questionnaire (NEQ) | at 5 weeks and at 6 months
  Monitoring and Reporting Adverse and Unwanted Events (32 items). Range 0-128 where a higher value indicates more adverse events.
Patient Health Questionnaire (PHQ-4) | Change from baseline health (PHQ-4) at 5 weeks
  Measures depressive symptoms and anxiety. Range 0-12 where a higher value indicates more depressive or anxiety symptoms.

CONTACTS AND LOCATIONS:
Overall Officials: Björn Gerdle, MD, PhD, Principal Investigator — Rehabilitation medicine, IMH, Linköping University
Locations (1):
- Rehabilitation medicine, IMH, Linköping University, Linköping, Östergötland County, Sweden

REFERENCES:
- [Derived] Wiklund T, Molander P, Lindner P, Andersson G, Gerdle B, Dragioti E. Internet-Delivered Cognitive Behavioral Therapy for Insomnia Comorbid With Chronic Pain: Randomized Controlled Trial. J Med Internet Res. 2022 Apr 29;24(4):e29258. doi: 10.2196/29258. PMID 35486418